CLINICAL TRIAL: NCT02541903
Title: A Phase 2 Trial Using Gilotrif for Advanced Penile Squamous Cell Carcinoma Following Systemic Therapy
Brief Title: Trial Using Gilotrif for Advanced Penile Squamous Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor overall accrual
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Lisle Nabell, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F150330009 (UAB 14113)
Record Dates: First submitted 2015-08-24; First posted 2015-09-04 (Estimated); Results first posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Penile Squamous Cell Carcinoma (PSCC)
Keywords: Epidermal growth factor receptor (EGFR),; Human Papillomavirus (HPV); Penile squamous cell carcinoma (PSCC); Gilotrif
MeSH Terms: interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gilotrif (Experimental): Gilotrif will be administered orally at 40 mg dosage once daily. Continuous administration of 4 weeks is considered one cycle. Therapy will continue until progression of the disease or severe toxicities. Labs will be monitored with routine blood collections every cycle and a CT scan will be done every two cycles (8 weeks).
  Interventions: Drug: Gilotrif

INTERVENTIONS:
Drug: Gilotrif — Patients will take a single oral dose of Gilotrif each day starting at 40 mg. Dose escalation and reductions can occur.

SUMMARY:
Penile squamous cell carcinoma (PSCC) is a highly aggressive and relatively rare disease. Supportive evidence for the value of systemic therapy does not exist for this disease and there are no agents currently approved by regulatory agencies. This study will evaluate the drug Gilotrif in patients with metastatic progressive PSCC following chemotherapy. Gilotrif has shown supportive evidence in non-small cell lung cancer by inhibiting certain proteins that are also found in PSCC. The drug has the potential for some patients to exhibit a response contributing to a greater quality of life.

DETAILED DESCRIPTION:
This is a non-randomized trial phase 2 trial in which the drug Gilotrif will be administered at an oral dosage of 40 mg daily. This will continue until there is disease progression or severe toxicities. Patients will undergo a clinical exam every 4 weeks as well as have blood collected. Radiographic scans will be done every 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed PSCC.
2. Patients with metastatic or locally advanced unresectable PSCC.
3. Progressive disease after ≥1 prior chemotherapy regimens.
4. Measurable disease by RECIST 1.1 criteria.
5. Prior regimen within 6 months
6. ECOG performance status 0-2.
7. Adequate organ function, defined as all of the following:

   * Absolute neutrophil count (ANC) >1500 /mm3. Platelet count >100,000/ mm3.
   * Estimated creatinine clearance ≥ 45ml/min.
   * Total Bilirubin <1.5 times upper limit of institutional normal; Aspartate amino transferase (AST) or alanine amino transferase (ALT) <2.5 times the upper limit of institutional normal (ULN).
   * Hemoglobin ≥8.5 g/dl.
8. Resolution of all acute toxic effects of prior chemotherapy or surgical procedures to NCI CTCAE version 4.03 grade <1, in the opinion of the Treating Physician.
9. Ability to understand and willingness to sign a written informed consent. Age ≥18 years or age of majority at the participating site, whichever is greater.
10. Availability of 20 archival formalin-fixed paraffin embedded tumor tissue slides.

Exclusion Criteria:

1. Patients will have recovered from toxicities from prior systemic anticancer treatment or local therapies.
2. Prior EGFR inhibitors.
3. Major surgery within 4 weeks or minor surgery within 2 weeks before registration or scheduled for surgery during the projected course of the study. Wounds will be completely healed prior to study entry and patients recovered from all toxicities from surgery. Placement of vascular access device is not considered major or minor surgery in this regard.
4. Prior radiation therapy is allowed as long as the irradiated area was not the sole source of measurable disease and radiotherapy was completed with recovery from toxicity, at least 3 weeks prior to enrollment. If the irradiated area is the only site of disease, there will be progressive disease.
5. History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure New York Heart Association (NYHA) classification of 3, unstable angina or poorly controlled arrhythmia as determined by the investigator. Myocardial infarction within 6 months prior to registration.
6. Any history of or concomitant condition that, in the opinion of the Investigator, would compromise the patient's ability to comply with the study or interfere with the evaluation of the efficacy and safety of the test drug.
7. Previous or concomitant malignancies at other sites, except effectively treated non-melanoma skin cancers, ductal carcinoma in situ or effectively treated malignancy that has been in remission for more than 3 years and is considered to be cured.
8. Requiring treatment with any of the prohibited concomitant medications listed in the protocol that cannot be stopped for the duration of trial participation.
9. Known pre-existing interstitial lung disease.
10. Any history or presence of poorly controlled gastrointestinal disorders that could affect the absorption of the study drug (e.g. Crohn's disease, ulcerative colitis, chronic diarrhea, malabsorption).
11. Active hepatitis B infection (defined as presence of Hep BsAg and/ or Hep B DNA), active hepatitis C infection (defined as presence of Hep C RNA) and/or known HIV carrier.
12. Meningeal carcinomatosis.
13. Patients with active brain or subdural metastases are not eligible, unless they have completed local (radiation) therapy and have discontinued the use of corticosteroids or have been on stable dose of corticosteroids for at least 4 weeks before starting study treatment. Any symptoms attributed to brain metastases will be stable for at least 4 weeks before starting study treatment.
14. Any active or uncontrolled infection.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-10; Primary Completion 2019-01-26 (Actual); Study Completion 2020-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisle Nabell, MD, Principal Investigator — University of Alabama at Birmingham; Tanya Dorff, MD, Study Chair — University of Southern California
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Southern California, Los Angeles, California
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was open to accrual between 10/6/2015 and 2/26/2019. Two sites were involved - the University of Alabama at Birmingham, and the University of Southern California.
Period: Overall Study
Arm/Group | Gilotrif
Started | 8
Completed | 7
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: 1 patient expired after signing consent but before starting treatment
Arm/Group | Gilotrif
Number analyzed (Participants) | 8
Age, Continuous [Mean (Full Range); unit: years] | 52.4 [33 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression Free Survival at 6 Months
Description: Death will signify the time of progression free survival. Otherwise, the Response Evaluation Criteria in Solid Tumors (RECIST) guidelines version 1.1 will be used to evaluate disease progression. Progression is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 6 months following study treatment
Population: 1 participant expired before receiving treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Gilotrif
Number analyzed (Participants) | 7
Participants | 1

2. Secondary Outcome: Response Rate
Description: The Response Evaluation Criteria in Solid Tumors guidelines version 1.1 and disease assessment scans (bone, CT) will be used to evaluate tumor response.
Time Frame: Baseline up to 3 months
Population: The response rate was calculated using those participants that showed regression or shrinkage at restaging scans.
Measure: Count of Participants; unit: Participants
Arm/Group | Gilotrif
Number analyzed (Participants) | 8
Participants | 2

3. Secondary Outcome: Overall Survival
Description: From date of study enrollment until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 30 months.
Time Frame: Baseline to death (assessed up to 30 months).
Measure: Mean (90% Confidence Interval); unit: days
Arm/Group | Gilotrif
Number analyzed (Participants) | 8
days | 83 [82 to 95]

4. Secondary Outcome: Toxicities
Description: The number of adverse events and serious adverse events will be tabulated using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: Baseline up to 18 months
Measure: Number; unit: Number of toxicities seen in patients
Arm/Group | Gilotrif
Number analyzed (Participants) | 8
Number of toxicities seen in patients | 5

ADVERSE EVENTS:
Time Frame: Adverse were collected every month during the study period and post-treatment (within 30 days)
Arm/Group | Gilotrif
All-Cause Mortality (participants affected / at risk) | 4/8
Serious Adverse Events (participants affected / at risk) | 4/8
Other Adverse Events (participants affected / at risk) | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gilotrif (N=8)
Fatigue (General disorders) | 1 (1) — Grade 2 fatigue requiring hospitalization
Death (General disorders) | 1 (1) — Patient died on C1D1 before starting treatment
Deep Venous Thrombosis (Vascular disorders) | 1 (1) — Grade 3
Hospitalization (Infections and infestations) | 1 (1) — Was admitted to the hospital for new drainage from L inguinal mass on 8/12/2017 , treated with Vanco/Zosyn and hyration. was given diaudid and norco for pain PRN. was discharged home on 8/15/2017
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gilotrif (N=8)
Decreased platelet count (Vascular disorders) | 1 (1)
cellulitis (Infections and infestations) | 1 (1)
Pain in scrotal region (General disorders) | 1 (1)
Anemia (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was closed early due to poor enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/03/NCT02541903/Prot_SAP_ICF_000.pdf